CLINICAL TRIAL: NCT04533620
Title: Predictive-Model Based Individualized Carbon-Ion Radiotherapy for Patients With Locally Recurrent Nasopharyngeal Carcinoma: A Phase 2 Randomized Trial
Brief Title: Individualized Carbon-Ion Radiotherapy for Patients With Locally Recurrent Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Jiade J. Lu, Prof. Jiade J. Lu, Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2020-46
Record Dates: First submitted 2020-08-24; First posted 2020-08-31 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Locally Recurrent Nasopharyngeal Carcinoma
Keywords: Locally recurrent nasopharyngeal carcinoma; Individualized carbon-ion radiotherapy; Predictive model of mucosal necrosis; Survival; Toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized CIRT (Active Comparator): Patients will receive standardized CIRT with a dose of 63 GyE/21 fx.
  Interventions: Radiation: Standardized CIRT
- Individualized CIRT (Experimental): A previously predictive model will be used to predict the chance of developing mucosal necrosis after salvage carbon-ion radiotherapy, and individualized dose prescription will be given. A dose of 60 GyE/20 fx, 63 GyE/21 fx and 66 GyE/22 fx will be given to patients with high, moderate and low risk of developing mucosal necrosis, respectively.
  Interventions: Radiation: Individualized CIRT

INTERVENTIONS:
Radiation: Standardized CIRT — CIRT with a dose of 63 GyE/21 fx
  Arms: Standardized CIRT
Radiation: Individualized CIRT — A predictive model will be used to predict the chance of developing mucosal necrosis after salvage carbon-ion radiotherapy, and individualized dose prescription will be given. A dose of 60 GyE/20 fx, 63 GyE/21 fx and 66 GyE/22 fx will be given to patients with high, moderate and low risk of developing mucosal necrosis, respectively.
  Arms: Individualized CIRT

SUMMARY:
This is a randomized phase 2 trial with 2 groups (control group vs experimental group). Patients with locally recurrent nasopharyngeal carcinoma (LR-NPC) assigned to the control group will receive standardized carbon-ion radiotherapy (CIRT). For patients assigned to the experimental group, a predictive model will be used to predict the chance of developing mucosal necrosis after salvage carbon-ion radiotherapy, and individualized dose prescription will be given. The primary endpoint of the study is to compare the 2-year progression-free survival (PFS) between 2 groups.

DETAILED DESCRIPTION:
This is a randomized phase 2 trial with 2 groups (control group vs experimental group). Patients with locally recurrent nasopharyngeal carcinoma (LR-NPC) assigned to the control group will receive standardized CIRT with a dose of 63 gray equivalent (GyE) in 21 fractions (fx). This regimen was obtained from our previous phase 1 (dose escalation) study. For patients assigned to the experimental group, a predictive model will be used to predict the chance of developing mucosal necrosis after salvage carbon-ion radiotherapy, and individualized dose prescription will be given. A dose of 60 GyE/20 fx, 63 GyE/21 fx and 66 GyE/22 fx will be given to patients with high, moderate and low risk of developing mucosal necrosis, respectively. The primary endpoint of the study is to compare the 2-year progression-free survival (PFS) between 2 groups. The secondary endpoints include 2-year overall survival (OS), local progression-free survival, regional progression-free survival, distant metastasis-free survival, toxicities and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 17-70 years.
* Pathologically diagnosed as WHO type 2/3 nasopharyngeal carcinoma.
* Failed previous definitive radiotherapy at least 6 months ago.
* Only had 1 previous course of radiotherapy.
* Eastern Cooperative Oncology Group score: 0-1.
* Adequate laboratory values within 30 dyas of enrollment to study defined as follows: 1) neutrophil > 2000/mm^3; 2) platelet > 100,000/mm^3; 3) total bilirubin < 1.5mg/dl; 4) alanine aminotransferase/aspartate aminotransferase < 1.5 upper limit of normal; 5) SCr < 1.5mg/dl; creatinine clearance rate > 60ml/min.
* Willing to accept adequate contraception for women with childbearing potential.
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial.

Exclusion Criteria:

* Presence of distant metastasis.
* Without measurable lesion.
* Previous history of malignant tumor (within 5 years) or simultaneous existence of multiple primary tumors.
* Accompanied with severe major organ dysfunction.
* Presence of mental disease that may influence the understanding of informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From randomization to death or disease progression, a median of 2 years

SECONDARY OUTCOMES:
Overall survival | From randomization to death, a median of 2 years
Local progression-free survival | From randomization to local failure, a median of 2 years
Regional progression-free survival | From randomization to regional failure, a median of 2 years
Distant metastasis-free survival | From randomization to distant metastasis, a median of 2 years
Incidence of radiation-induced acute toxicity evaluated by CTCAE 5.0 | Within 3 months after initiation of radiation therapy
Incidence of radiation-induced late toxicity evaluated by CTCAE 5.0 | Three months after initiation of radiation therapy
Quality of life by questionnaires evaluated using EORTC-Q30 questionnaire. | Throughout the study, an average of 2 years
Quality of life by questionnaires evaluated using EORTC-H&N35 questionnaire. | Throughout the study, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jiade J Lu, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including baseline characteristics, treatment information and follow-up data on toxicity, survival and disease control will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within 5 years after the publication of the study.
Access Criteria: Data may be shared with radiation oncologists who are interested in examining the efficacy and toxicity of locally recurrent nasopharyngeal carcinoma patients treated with particle beam radiotherapy. Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.